CLINICAL TRIAL: NCT00139087
Title: Mother-Infant Rapid Intervention at Delivery Telephone Outreach for Neonatal Therapy (TOT) Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3010
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2005-08-31 (Estimated); Status verified 2005-08

CONDITIONS: HIV
MeSH Terms: interventions — Therapeutics

INTERVENTIONS:
Behavioral: Telephone Outreach for Therapy

SUMMARY:
The Telephone Outreach for Therapy Trial was designed to test an intervention to assist new mothers or caregivers of HIV-exposed children with administering medication for the first 6 weeks of life to prevent mother-to-child HIV infection in the infants. To be eligible, mothers of infants were identified as HIV-infected in the Mother-Infant Rapid Intervention at Delivery Study. Mothers or caregivers of infants were randomized into two groups: the intervention group received a cellular phone and scheduled twice daily calls to assure infant medications were given, and the other group received the current standard of care. Enrollment into the study was completed and analysis of the study data is underway.

DETAILED DESCRIPTION:
The Telephone Outreach for Therapy Trial was designed to test an intervention to assist new mothers or caregivers of HIV-exposed children with administering medication for the first 6 weeks of life to prevent mother-to-child HIV infection in the infants. To be eligible, mothers of infants were identified as HIV-infected in the Mother-Infant Rapid Intervention at Delivery Study. Mothers or caregivers of infants were randomized into two groups: the intervention group received a cellular phone and scheduled twice daily calls to assure infant medications were given, and the other group received the current standard of care. Enrollment into the study was completed and analysis of the study data is underway.

ELIGIBILITY:
Inclusion Criteria:

* Mother-infant pairs in which the mother was identified as HIV-infected in the MIRIAD Study

Exclusion Criteria:

* Mother-infant pairs in which the infant is expected to be hospitalized for >2weeks after birth

Ages: 1 Hour to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300
Dates: Start 2002-01; Study Completion 2005-03

PRIMARY OUTCOMES:
Neonatal adherence to zidovudine syrup measured as self report of the mother or caregiver AND drug level measured in heel stick specimens collected at 2, 4 and 6 weeks of life.

CONTACTS AND LOCATIONS:
Overall Officials: Susan P Danner, BA, Study Director — Centers for Disease Control and Prevention